CLINICAL TRIAL: NCT04297995
Title: Evaluate the Efficacy and Safety of HLX10, PD-1 mAb, in Combination With HLX07, EGFR mAb, in Patients With Advanced Head And Neck Tumors
Brief Title: Evaluate the Efficacy and Safety of HLX10 in Combination With HLX07 in Patients With Advanced Head and Neck Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HLX10HLX07-001
Record Dates: First submitted 2020-03-02; First posted 2020-03-06 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — HLX07; Cisplatin; Carboplatin; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Part 1: open label.
  Part 2: Matters related to the blinding of study treatment will be carried out by the statistics department. The subjects, the INV, the sponsor, and designees are not aware of the randomized allocation. This study will be unblinded overall approximately 3 months after the first administration in the last subject. Unblinding is allowed unless there is an emergency medical condition (emergency treatment is only possible when being informed of the randomized medication) or unblinding is requested by the regulatory authorities. Otherwise, the study should remain blinded. Only when all data have been input into the database, all data queries have been resolved, and subjects have been allocated into analysis sets, can the randomization codes be unblinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1: HLX10 Plus HLX07 (stage 1L) (Experimental): 3 mg/kg of HLX10 every two weeks infusion combined with 600 mg HLX07 weekly
  Interventions: Drug: HLX10; Drug: HLX07
- Part 1: HLX10 Plus HLX07 (Stage 1H) (Experimental): 3 mg/kg of HLX10 every two weeks infusion combined with 800 mg HLX07 weekly
  Interventions: Drug: HLX10; Drug: HLX07
- Part 2: HLX10 Plus HLX07 Plus Chemotherapy (Experimental): HLX10 (300 mg) Plus HLX07 (1000 mg) Plus Cisplatin (100 mg/m2) Plus 5-FU (1000 mg/m2/day, 1-4 days). Cisplatin will be switched to carboplatin in case of intolerance to cisplatin. Up to 6 cycles of chemotherapy.
  Interventions: Drug: HLX10; Drug: HLX07; Drug: Cisplatin/Carboplatin; Drug: 5-FU
- Part 2: HLX10 Plus HLX07 Placebo Plus Chemotherapy (Placebo Comparator): HLX10 (300 mg) Plus HLX07 Placebo (1000 mg) Plus Cisplatin (100 mg/m2) Plus 5-FU (1000 mg/m2/day, 1-4 days). Cisplatin will be switched to carboplatin in case of intolerance to cisplatin. Up to 6 cycles of chemotherapy.
  Interventions: Drug: HLX10; Drug: HLX07 placebo; Drug: Cisplatin/Carboplatin; Drug: 5-FU

INTERVENTIONS:
Drug: HLX10 — Part 1: HLX10 3 mg/kg biweekly. Part 2: HLX10 300 mg every three weeks.
Drug: HLX07 — Part 1: HLX07 600 mg weekly (stage 1L). Part 1: HLX07 800 mg weekly (stage 1H). Part 2: HLX07 1000 mg every three weeks.
  Arms: Part 1: HLX10 Plus HLX07 (Stage 1H); Part 1: HLX10 Plus HLX07 (stage 1L); Part 2: HLX10 Plus HLX07 Plus Chemotherapy
Drug: HLX07 placebo — HLX07 placebo 1000 mg every three weeks
  Arms: Part 2: HLX10 Plus HLX07 Placebo Plus Chemotherapy
Drug: Cisplatin/Carboplatin — Cisplatin 100 mg/m2 every three weeks. Cisplatin will be switched to carboplatin in case of intolerance to cisplatin. Up to 6 cycles.
  Arms: Part 2: HLX10 Plus HLX07 Placebo Plus Chemotherapy; Part 2: HLX10 Plus HLX07 Plus Chemotherapy
Drug: 5-FU — 5-FU 1000 mg/m2/day, 1-4 days, every three weeks. Up to 6 cycles.
  Arms: Part 2: HLX10 Plus HLX07 Placebo Plus Chemotherapy; Part 2: HLX10 Plus HLX07 Plus Chemotherapy

SUMMARY:
Part1:

A mutilpe-center, open-label, Phase II clinical trial to evaluate the efficacy and the safety of HLX10 in combination with HLX07 in patients with advanced advanced head and neck tumors.

Part2:

A randomized, double-blind, multi-center, phase II clinical study to evaluate the clinical efficacy and safety of HLX10 in combination with HLX07 and chemotherapy versus HLX10 in combination with placebo and chemotherapy in the first-line treatment of R/M HNSCC.

DETAILED DESCRIPTION:
Part 1:

This is an open label study. Sample size recommendations for this phase II study are determined according to Simon's two-stage Optimal design.

In the first stage, 13 patients will be accrued. The patients will receive 3 mg/kg of HLX10 every two weeks infusion combined with 600 mg HLX07 weekly (stage 1L). These patients will be assessed for treatment response after 8 weeks of first infusion of study drugs. If there are 3 or fewer responsive patients in these 13 patients, additional 13 patients will be accrued. These additional 13 patients will receive 3 mg/kg of HLX10 every two weeks infusion combined with 800 mg HLX07 weekly (Stage 1H). If 3 or fewer responses after eight weeks treatment noted in these 13 patients in stage 1H, the trial will be stopped.

If 4 or more patients are responsive to therapy in stage 1, the trial will be continued to stage 2, 30 additional patients will be accrued to reach a total of 43 patients. These additional 30 patients will receive the same dose of regimen as the prior patients.

Part 2:

This is a randomized, double-blind, multi-center, phase II clinical study to evaluate the clinical efficacy and safety of HLX10 in combination with HLX07 and chemotherapy versus HLX10 in combination with placebo and chemotherapy in the first-line treatment of R/M HNSCC. Approximately 75 first-line R/M HNSCC subjects are planned to be recruited. The sample size calculation is not based on the statistical hypothesis.

Eligible subjects after screening will be randomly assigned to the treatment group (group A) or the control group (group B) in a ratio of 2:1, with PD-L1 CPS (≥ 20 and < 20) as the stratification factor at randomization (Figure 1):

Group A: approximately 50 subjects, HLX10 in combination with HLX07 and chemotherapy (cisplatin in combination with 5-FU).

Group B: approximately 25 subjects, HLX10 in combination with placebo and chemotherapy (cisplatin in combination with 5-FU).

Cisplatin may be replaced with carboplatin when the subject is judged intolerant to cisplatin by the INV.

The study will be unblinded overall for ORR analysis approximately 3 months after the first dose of the last subject.

ELIGIBILITY:
Part1

Inclusion Criteria:

1. Eligible patients must be 18 years of age or older or per local regulation AND younger than 80 years old age.
2. Patients with histologically-proven recurrent (not amenable to locally curative treatment options) or metastatic, squamous cell carcinoma of the head and neck with previously failed platinum-based chemotherapy and PD-L1 expression (combined positive score ≥ 1) as determined by immunohistochemistry (IHC) stain. (Patient must be able to provide tissue for PD-L1 biomarker analysis from a core or excisional biopsy; fine needle aspirate is not sufficient.: A newly obtained biopsy; within 90 days prior to start of study treatment; is preferred but an archival sample is acceptable.)
3. Lesion must be measurable based on RECIST, version 1.1.
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1 at the time of study entry.
5. Able to provide informed consent.
6. A life expectancy longer than three months.
7. Adequate hematologic functions, as defined by: absolute neutrophil counts (ANC) ≥ 1500/mm3; a hemoglobin (Hb) level ≥ 9 gm/dL; a platelet count ≥ 100,000/mm3.
8. Adequate hepatic function defined by: a total bilirubin level ≤ 1.5x of upper limit of normal (ULN); aspartate transaminase (AST) and alanine transaminase (ALT) levels ≤ 2.5 x of ULN or ≤ 5x of ULN in known hepatic metastases.
9. Adequate renal function, as defined by the creatinine clearance rate ≥ 50 mL/minute calculated using Cockcroft-Gault formula. In patient with extreme body weight (body mass index [BMI] < 18.5 or > 30), estimated glomerular filtration rate (GFR) ≥ 50mL/min calculated using Modification of Diet in Renal Disease (MDRD) formula is acceptable.
10. Adequate cardiac function defined as left ventricular ejection fraction (LVEF) ≥ 50% measured by multigated acquisition (MUGA) scan or cardiac ultrasound.
11. Use of effective contraceptive measures if procreative potential exists .
12. At least 28 days from prior major surgery, prior cytotoxic chemotherapy, or prior therapy with investigational agents (or medical device) and curative radiotherapy or palliative radiotherapy to target lesion before the first infusion of investigational product.
13. Able to follow the procedures as required by the study protocol and must agree to provide tumor tissue for programmed cell death 1 (PD-L1) expression analyses, EGFR mutation status, and biomarker assessment.

Exclusion Criteria:

1. Patients who still have persistent ≥ grade 2 toxicities from prior therapies.
2. Patients with primary nasopharynx cancers.
3. Squamous cell carcinoma of unknown primary in cervical lymph node.
4. Concurrent unstable or uncontrolled medical conditions. Either of the followings:

   * Active systemic infections currently under treatment with antimicrobial agents;
   * Poorly controlled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥100 mmHg), or poor compliance with anti-hypertensive agents;
   * Clinically significant arrhythmia, unstable angina pectoris, congestive heart failure (class III or IV of New York Heart Association [NYHA]) or acute myocardial infarction within 12 months;
   * Uncontrolled diabetes or poor compliance with hypoglycemic agents;
   * The presence of chronically unhealed wound or ulcers;
   * Other chronic diseases, which, in the opinion of the investigator, could compromise safety of the patient or the integrity of study.
5. Newly-diagnosed or symptomatic brain metastases (patients with a history of brain metastases must have received definitive surgery or radiotherapy, must be clinically stable, and must not taking steroids for brain edema for at least 14 days to be allowed in the study). Anticonvulsants are allowed.
6. Any concurrent malignancy other than basal cell carcinoma or carcinoma in situ of the cervix. (Patients with a previous malignancy but without evidence of disease for ≥ 3 years can participate).
7. Pregnancy (confirmed by serum beta human chorionic gonadotropin [ßHCG]) or breast-feeding.
8. Known history of human immunodeficiency virus infection (HIV).
9. Patient who has an active or a documented history of autoimmune disease.
10. Patient who has active hepatitis B (HBV DNA titer > 100 IU/mL or > 500 copies/mL) or hepatitis C (defined as anti-HCV antibody reactive and/ or detectable HCV RNA > 15 IU/L).
11. Patient who has a history of interstitial lung disease.
12. Have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of autoimmune disease.
13. Patients who have failed systemic anti-EGFR monoclonal antibody therapies (who have PD or PFS less than 3 months during anti EGFR treatment) or have been received more than 3 lines of systemic chemotherapy regimens.
14. Patients who previously have severe allergic reaction to anti-EGFR monoclonal antibody (CTCAE grade ≥3).
15. Patients who have previously received immune check point therapy, including but not limit to anti-PD1 and anti-PDL1.
16. The patient is the investigator, sub-investigator or any one directly involved in the conduct of the study.
17. Patient has a history or current evidence of any condition or disease that could confound the results of the study, or study or is not the best interest of the patient to participate, in the opinion of Investigator.

Part2

Inclusion Criteria:

1. Histologically or cytologically confirmed R/M HNSCC that is considered incurable by local therapies.
2. Have not received any systemic anti-tumor therapy for R/M HNSCC. Patients who have received systemic anti-tumor therapy (including anti-EGFR antibody drugs) as part of comprehensive treatment at the locally advanced stage are allowed to be enrolled if the systemic therapy has been completed for at least 6 months before signing the informed consent form (ICF).

   * Tumor types to be included: primary cancers of the oropharynx, oral cavity, hypopharynx, and larynx.
   * Patients with primary nasopharyngeal cancer are not allowed to be enrolled.
   * Willing and able to provide the written ICF to participate in this study.
3. Age ≥ 18 years at the time of signing the ICF.
4. Have measurable lesion as assessed by the INV per RECIST v1.1. Previously irradiated lesions may be considered measurable if progression has been confirmed in such lesions.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at the time of enrollment.
6. Normal major organ functions.
7. Able to provide tissue samples from needle biopsy or excisional biopsy (fine-needle aspiration is unacceptable) for determination of EGFR and PD-L1 expression. Patients with oropharyngeal cancer are required to provide additional tissue samples for HPV (P16) status testing. Tissue samples should be re-collected if the quantity is not adequate.
8. Female subjects with childbearing potential must be tested negative for serum pregnancy test within 7 days prior to the first dose.
9. Female subjects with childbearing potential should agree to use two methods of contraception, undergo sterilization, or avoid heterosexual sex during the treatment and until 180 days after the last dose. Subjects with childbearing potential refer to those who have not undergone sterilization or have stopped menstruating for less than 1 year. Subjects are allowed to choose abstinence as a contraceptive measure if abstinence is their normal lifestyle.
10. Male subjects should agree to take adequate contraceptive measures from the first dose until 180 days after the last dose. Subjects are allowed to choose abstinence as a contraceptive measure if abstinence is their normal lifestyle.

Exclusion Criteria:

1. Subjects who are candidates for radical locoregional therapy.
2. PD within 6 months after completion of radical systemic therapy (including anti-EGFR antibody drugs) for locally advanced HNSCC.
3. Have received radiotherapy (or other non-systemic therapies) within 2 weeks prior to the first dose or still have AEs related to previous treatment that have not fully recovered (e.g., to ≤ grade 1 or to baseline).

   * Subjects with ≤ grade 2 neuropathy, or ≤ grade 2 alopecia, or laboratory parameters meeting Article 6 of the inclusion criteria are not subject to this exclusion criterion and are allowed to be enrolled.
   * For subjects who have undergone major surgery, surgery-related toxicity or complications must be fully recovered before the first dose. The major surgery in this study is defined as a surgery requiring at least 3 weeks of recovery for a subject to be able to receive the treatment in this study.
4. Currently on other clinical study treatment, or have received treatment with other IPs or medical devices within 4 weeks prior to the first dose. Subjects who are in the follow-up period of the previous clinical study (not in the study treatment period) are allowed to be enrolled.
5. Life expectancy of less than 3 months and/or rapid disease progression (e.g., tumor bleeding, uncontrolled neoplastic pain) as judged by the INV.
6. Myocardial infarction or poorly controlled arrhythmia (including QTc intervals ≥ 450 ms for males and ≥ 470 ms for females) (QTc intervals are calculated by Fridericia's formula) within 6 months prior to the first dose.
7. Class III to IV cardiac insufficiency according to New York Heart Association (NYHA) classification or a left ventricular ejection fraction (LVEF) < 50% by cardiac color Doppler.
8. Subjects with inadequately controlled hypertension (systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 100 mmHg), showing a history of hypertensive crisis or hypertensive encephalopathy.
9. Artery/vein thrombosis or thromboembolism events, including pulmonary embolism, occurred within 6 months prior to the first dose.
10. Subjects who have a diagnosis of immunodeficiency or are receiving systemic steroid treatment or any other forms of immunosuppressive therapy within 7 days prior to the first dose. Corticosteroids can be used as prophylactic medications for anaphylaxis (e.g., intravenous contrast agent) or for prophylactic management of chemotherapy-related AEs as specified in the protocol. Corticosteroids at physiologic doses are allowed upon consultation with the sponsor.
11. Other malignancies diagnosed and/or treated within 3 years prior to the first dose with the exception of: curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, radically resected cervical carcinoma in situ, and radically resected breast cancer in situ. Other exceptions may be considered in consultation with the sponsor.
12. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Note: Subjects with previously treated brain metastases may participate in this study when meeting the following criteria: stable condition for at least 4 weeks prior to the first dose (showing no imaging evidence of progression (under the same imaging mode for each evaluation, either MRI or CT scan), with all neurological symptoms back to baseline); no evidence of new or expanded brain metastases; no use of steroids within at least 7 days prior to the first dose. Carcinomatous meningitis should be excluded regardless of clinical stability.
13. Active autoimmune disease requiring systemic therapy (e.g., disease-modifying drugs, corticosteroids, or immunosuppressants) present within 2 years prior to the first dose. Alternative therapies (e.g., thyroxine, insulin, or physiologic corticosteroids for adrenal or pituitary insufficiency) are not considered systemic therapies.
14. Have received transplantation of allogeneic tissues or parenchymal organs.
15. A history of previous or current pneumonitis (non-infectious) requiring steroid therapy.
16. Active infection requiring systemic therapy.
17. Subjects whose medical history or current abnormal laboratory data may cause confusion about study results or interference in their full participation in this study, or for whom participation in this study is not in their best interest as assessed by the INV.
18. Known mental disorders or drug abuse that will interfere with the subject's compliance with the requirements of this study.
19. Pregnant or lactating women, or those who prepare to become pregnant or give birth during the expected duration of this study (from the screening visit to 180 days after the last dose).
20. Patients who have been treated with immune checkpoint inhibitors (including but not limited to anti-PD-1 or anti-PD-L1 antibody drugs).
21. Known history of human immunodeficiency virus (HIV) infection.
22. Positive (+) for hepatitis B surface antigen (HBsAg) or positive (+) for hepatitis B core antibody (HBcAb), and with hepatitis B virus deoxyribonucleic acid (HBV-DNA) ≥ 2500 copies/mL or 500 IU/mL, or presence of active hepatitis determined clinically (patients whose HBV-DNA has decreased below the above criteria after antiviral therapy and who are willing to receive antiviral therapy throughout the study are allowed to be enrolled); patients with hepatitis C (positive for HCV-RNA).
23. Have received live vaccines within 30 days prior to the first dose.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Part1: Efficacy-ORR | at 16 weeks after first dose
  Objective Response Rate (ORR)
Part1: Safety-adverse event profile | up to one year
  The proportion of patients suffered from drug related toxicities.
Part2: Efficacy-ORR (IRRC) | at 3 months after first dose
  Objective Response Rate (ORR) assessed by the Independent Radiological Review Committee (IRRC) per RECIST v1.1.

SECONDARY OUTCOMES:
Efficacy-Best ORR | up to one year
  Best response rate (Best ORR)
Efficacy-PFS | up to one year
  Progression-free survival (PFS)
Efficacy-OS | up to one year
  Overall survival (OS)
The number of presence patients that develop of anti-durg antibody (immunogenicity). | up to one year
maximum concentration (Cmax) | up to one year
trough concentration (Ctrough) | up to one year
half-life (T1/2) | up to one year
clearance rate (CL) | up to one year
volume of distribution (Vss) | up to one year
area under concentration (AUC0-tau) | up to one year

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, PhD, Principal Investigator — Shanghai East Hospital; Guochun Cao, Principal Investigator — Jiangsu Cancer Institute & Hospital; Meiyu Fang, Principal Investigator — Cancer Hospital of The University of Chinese Academy of Sciences; Guangyuan Hu, Principal Investigator — Tongji Hospital; Xiaohui He, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Yan Sun, Principal Investigator — Peking University Cancer Hospital & Institute; Wei Wang, Principal Investigator — Hunan Cancer Hospital; Shubin Wang, Principal Investigator — Peking University Shenzhen Hospital; Qingyuan Zhang, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (1):
- Shanghai Henlius Biotech Inc., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Y. Guo, W. Wang, G. Cao, et al. A phase 2 study of serplulimab plus HLX07 in patients with advanced head and neck tumours. Abstract Book. ICHNO-ECHNO 2022: 590
- [Derived] Wang K, Shen Y, Hu C, Xu F, Wang Q, Gao Y, Zhou L. Population Pharmacokinetics and Exposure-Response Analysis of Serplulimab in Small Cell Lung Cancer Patients. Clin Transl Sci. 2025 Sep;18(9):e70322. doi: 10.1111/cts.70322. PMID 40932107
- See also: Related Info — http://user-swndwmf.cld.bz/ICHNO-ECHNO-2022-Abstract-Book/100/